CLINICAL TRIAL: NCT02694289
Title: Effects of Metformin in Heart Failure Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: failure to enroll participants
Sponsor: Maya Guglin (Other)
Responsible Party: Sponsor-Investigator, Maya Guglin, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-0797-F6A
Record Dates: First submitted 2016-02-05; First posted 2016-02-29 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Injections, Subcutaneous; Insulin; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Other): Continue Metformin while admitted to hospital
  Interventions: Drug: Metformin
- Subcutaneous (sliding scale) Insulin (Other): Discontinue Metformin upon admission and be placed on sliding scale subcutaneous insulin treatment while admitted to hospital
  Interventions: Drug: Subcutaneous (sliding scale) Insulin

INTERVENTIONS:
Drug: Metformin — Treatment/continuation of metformin therapy during admission
  Other Names: no other names
  Arms: Metformin
Drug: Subcutaneous (sliding scale) Insulin — Discontinue Metformin and be placed on subcutaneous sliding scale insulin during admission
  Other Names: eg. Humulin, Lantus, Novalin
  Arms: Subcutaneous (sliding scale) Insulin

SUMMARY:
Hypothesis: In patients, who have diabetes type 2, are treated with metformin, and are admitted for HF, leads to reduced insulin requirements, as measured in units of insulin, with no negative impact on patient safety.

This is a single center, prospective trial. Subjects will be randomized to initiate metformin (starting dose 500mg orally once daily up to a maximum dose of 2,500mg daily) OR be placed on insulin products for management of their type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Because of the state of insulin resistance in heart failure (HF), metformin, with its ability to sensitize tissues to insulin, seems to be an ideal agent for managing type 2 diabetes mellitus (DM) in HF. It reduces the concentration of glucose in blood by enhancing insulin sensitivity, inducing greater peripheral uptake of glucose, and decreasing hepatic glucose output. However, according to the package insert, it is contraindicated in all patients with HF requiring pharmacologic treatment because of increased risk of lactic acidosis. The FDA has now de-escalated this contraindication to a warning as the evidence is lacking regarding an increased risk of lactic acidosis in patients with type 2 DM and HF who take metformin.

Hypothesis: In patients, who have diabetes type 2, are treated with metformin, and are admitted for HF, metformin leads to reduced insulin requirements, as measured in units of insulin, with no negative impact on patient safety.

Primary Objective: To test the hypothesis that continuing a patient's home metformin for diabetes management while admitted to UK hospital will result in decreased utilization of insulin as denoted by total units given.

Secondary Objectives: To test the hypothesis that administering metformin in HF patients admitted to UK Hospital:

1. Results in similar glycemic control (targeting a blood glucose < 200mg/dL) when compared with placebo along on the basis of basic metabolic panel glucose values. Both groups may receive conventional inpatient hyperglycemia management with insulin products
2. Reduces drug and laboratory costs
3. Reduces hospital length of stay
4. Does not result in hypoglycemia (blood glucose < 60 mg/dL)
5. Reduced discharge medication errors related to diabetic medications
6. No observed increase in metabolic acidosis due to elevated lactate levels
7. Does not impact heart failure status (as indicated by trending NT-pro BNP levels)

Both the diagnosis and clinical management of patients with heart failure and type 2 diabetes mellitus will be guaranteed by the application of standard guidelines internationally recognized. All patients admitted to the Medicine / Cardiology Advanced Heart Failure at UK Hospital will be evaluated for inclusion and exclusion criteria. Based on our power analysis we plan to enroll 100 subjects total. Subjects will be enrolled from January 1, 2016 - December 31, 2018 until 120 patients are enrolled, estimated study time frame is two years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > / = 18 years of age
2. Admitted to the Medicine / Cardiology Advanced Heart Failure at UK Hospital
3. Carry a diagnosis of heart failure with or without preserved ejection fraction
4. Carry a diagnosis of type 2 diabetes mellitus

Exclusion Criteria:

1. Patients <18 years of age
2. Prisoners
3. Terminal state
4. Known adverse reaction or hypersensitivity to metformin administration
5. Pregnancy
6. Pathological conditions in which metformin administration is clinically contraindicated (Patients with acute or chronic metabolic acidosis, serum creatinine > 1.4 mg/dL in females, serum creatinine > 1.5 mg/dL in males)
7. Patients with acute cardiovascular collapse, acute myocardial infarction, septicemia
8. Patients carrying a diagnosis of type 1 diabetes mellitus
9. Patients admitted with diabetic ketoacidosis or hyperosmotic hyperosmolar state.
10. Patients who experience diabetic ketoacidosis or hyperosmotic hyperosmolar state at any point during their hospital admission.
11. Patients admitted with a subcutaneous insulin pump
12. Patients who, at the discretion of the Medicine / Cardiology Advanced Heart Failure service, required an endocrinology consult during their hospitalization where the endocrine consult service is opposed to utilizing metformin in a particular patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Units of Insulin used | from time of hospital admission to hospital discharge, up to one year
  doses and amounts on insulin needed

SECONDARY OUTCOMES:
Blood glucose levels | from time of hospital admission to hospital discharge, up to one year
  patient's glycemic control will be evaluated based on blood glucose levels
Length of stay | time from hospital admission to hospital discharge, up to one year
Lactate levels, mmol/L | from time of hospital admission to hospital discharge, up to one year
pro-BNP levels, pg/mL | from time of hospital admission to hospital discharge, up to one year

CONTACTS AND LOCATIONS:
Overall Officials: Maya Guglin, MD, PhD, Principal Investigator — University of Kentucky

IPD SHARING:
Plan to Share IPD: No